CLINICAL TRIAL: NCT07137221
Title: Acupunture And Inflammatory Status In Breast Cancer Patients With Climateric Syndrome: A Pilot Study (FLAIR: Flushes, Acupuncture, Inflammation Research)
Brief Title: Acupuncture And Inflammatory Status In Breast Cancer Patients With Climateric Syndrome.
Acronym: FLAIR
Status: Completed | Type: Observational
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: IRSTB104
Record Dates: First submitted 2025-08-06; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Observational; postmonopausal; breast cancer; Hot Flashes; Acupuncture; Adjuvant Therapy; Prospective Study; Inflammation
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh peripheral bloodsamples will be collected at baseline, after 10 weeks and after 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post menopausal breast cancer patients: Prospective cohort.
  Interventions: Other: Post menopausal breast cancer patients

INTERVENTIONS:
Other: Post menopausal breast cancer patients — All selected patients will undergo peripheral blood samplingfor the evaluation of inflammatory biomarkers and must have agreed to store and use part of their sample for research purposes.
  A panel of inflammatory cytokines (IFNγ, IL-1β, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12p70, IL-22, TNFα) will be detected by ELISA assay. Other biomarkers such as RANKL, OPG, Vitamin D levels, CTX, PTH will be evaluated by immunoenzymatic assays. In addition, mirNAs as mir-16 and mir-378 will be evaluated by RT-PCR. Glucose metabolic markers such as fasting glucose and insulin, HbA1c and other parameters such as calcemia, PTH, c-telopeptide etc. will be collected.
  In particular, the evaluation of the biomarkers will be done on plasma samples at different time points (previously the administration of 10 course of weekly acupuncture; at the end and 6 months after the end of acupuncture and at the time of symptoms recurrence.

SUMMARY:
This is a prospective, single-center, non-interventional, non-pharmacological study.

In this study, postmenopausal patients with breast cancer in the adjuvant setting will be enrolled and treated with acupuncture to reduce hot flashes and other climacteric symptoms.

DETAILED DESCRIPTION:
In healthy postmenopausal women, hot flashes (HF) have been associated with systemic inflammation.

Several studies suggest that acupuncture (ACU) is effective in improving menopausal HF symptoms, both in healthy women and in patients with breast cancer. The effectiveness of ACU appears to be independent of changes in estradiol, FSH, and LH levels; however, the precise mechanisms through which ACU alleviates HF have not yet been clearly documented.

Various studies indicate that menopause may trigger an increase in pro-inflammatory cytokines, likely due to the decline in sex hormone levels. Moreover, the elevated levels of pro-inflammatory factors during menopause may be linked to later health events, such as the development of osteoporosis and atherosclerosis.

The literature highlights a connection between increased activity of pro-inflammatory cytokines-particularly IL-6-and postmenopausal bone loss, involving the RANK and Osteoprotegerin (OPG) pathways.

The severity of HF is also significantly associated with the HOMA index and other markers of insulin resistance. This suggests a possible correlation between the severity of postmenopausal HF and the risk of cardiovascular disease, including in breast cancer patients.

The primary objective of this study is to investigate the biochemical mechanisms underlying the effectiveness of acupuncture in alleviating hot flashes and other climacteric symptoms in postmenopausal women with breast cancer. Specifically, the study aims to determine whether the clinical benefits observed with acupuncture treatment are associated with measurable changes in inflammatory dysregulation in this patient population.

In addition to the primary objective, the study includes several secondary aims. These involve evaluating the relationship between the improvement of postmenopausal symptoms and various biological markers, including indicators of bone loss, insulin resistance, hormone levels, and lipid profile. Furthermore, the study seeks to explore the correlation between circulating biomarkers and pain relief, as measured through validated instruments such as the EQ-5D-5L and BPI questionnaires, in the context of acupuncture treatment.

It is anticipated that approximately 60 patients will participate, and the study will last a total of 42 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a previous diagnosis of breast cancer.
* Not metastatic disease
* Disorders of thermoregulation with or without any other symptoms referable to the syndrome menopausal or perimenopausal from at least 6-8 weeks prior study entry
* Age 18-65 years
* patients with postmenopausal breast cancer defined as follows:

  * bilateral oophorectomy
  * age ≥ 60 years
  * age ≤ 60 years, who has had at least 12 consecutive months of amenorrhea in the absence of any adjuvant treatment and serum dosage of FSH and E2 in the postmenopausal range (FSH> 40IU/L and E2 <10 pg/ml)
  * age <60 years, treated with tamoxifen or aromatase inhibitors and serum dosage of FSH and E2 in the postmenopausal range (FSH> 40UI/L and E2 <10 pg/ml)
  * patients treated with GhRh analogues for at least 3 months in combination with tamoxifen or aromatase inhibitors for at least 2 months .- Early Postmenopause stage (≤ 5 years) based on Stages of Reproductive Aging Workshop (STRAW) criteria
* BMI within the range of ≥18.5 Kg/m² and less than 24.5 kg/m²
* Number of hot flushes greater than or equal to an average of 6/day in the week and / or average daily score on the climacteric scale of Greene> of 15 prior to enrolled in study
* ECOG performance status < or equal to 1
* Not previous diagnosis of inflammatory disorders such as rheumatic, respiratory, dermatologic, no gastroenterologic acute and chronic diseases; none immunological altered condition; no type 1 and 2 diabetes, hypertension, hyperlipidemia; no thyroid diseases or neurodegenerative diseases;
* not women smokers
* not concomitant homeopaty or phytotherapy treatment, corticosteroid, NSAID, antidepressant drugs
* written informed consent

Exclusion Criteria:

* Age < 18 or > 65 years
* Metastatic breast cancer
* Previous diagnosis of inflammatory disorders such as rheumatic, respiratory, dermatologic, gastroenterologic acute and chronic diseases; any immunological altered condition; type 1 and 2 diabetes; uncontrolled hypertension; hyperlipidemia in treatment; autoimmune thyroid diseases; neurodegenerative diseases;
* smoker;
* Concomitant homeopathy or phytotherapy treatment, corticosteroid, NSAID, antidepressant drugs
* Language or educational barriers to understanding the study purpose

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Disorders of thermoregulation with or without any other symptoms referable to the syndrome menopausal or perimenopausal from at least 6-8 weeks prior study entry.
Study Population: Post menopausal breast cancer patients, it is expected that 60 patients may participate.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Acupuncture Effects on Inflammation and Menopausal Symptoms in Breast Cancer | 42 months
  Change in Greene Climacteric Scale evaluated before (T0) and after treatment (ten weeks of treatment (T1) and six-month follow-up (T2)). The scale assigns a rating to the disruption caused by each symptom, ranging from 0 (undisturbed) to 3 (extremely disturbed), across three symptom categories: psychological, physical, and vasomotor. These categories are defined by 21 items, with a total score that ranges from 0 to 63. The mean value of menopausal symptoms experienced over seven consecutive days will be calculated, and changes observed between baseline (T0) and after ten weeks of treatment (T1) and six-month follow-up (T2) will be documented.

SECONDARY OUTCOMES:
Correlation Between Symptom Improvement and Metabolic Markers in Postmenopausal Women. | 42 months
  Changes in hot flash intensity, inflammatory cytokine levels (IFN-γ, IL-1β, IL-4, IL-5, IL-6, IL-8, IL-10, IL-22, TNF-α), menopausal symptoms, markers of insulin resistance (fasting glucose, insulin, glycated hemoglobin), lipid profile (total cholesterol, HDL, LDL, triglycerides), bone density (calcium, vitamin D, parathyroid hormone, C-telopeptide), hormonal levels (FSH, LH, estradiol), quality of life (EQ-5D-5L questionnaire) and pain level (Brief Pain Inventory scale) evaluated before and after treatment.
Correlation of Biomarkers with Pain Relief and Acupuncture | 42 months
  Circulating markers with pain relief (EQ-5D-5L and BPI) questionnaires and acupuncture procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Fedeli, Dr., Study Director — IRCCS IRST
Locations (1):
- Irccs Irst, Meldola, FC, Italy

IPD SHARING:
Plan to Share IPD: No